CLINICAL TRIAL: NCT02443168
Title: A Phase 1, Open-Label, Two-Part Study to Evaluate the Metabolism, Excretion, and Absolute Bioavailability of AG-221 in Healthy Adult Male Subjects
Brief Title: Radiolabeled Study of AG-221 in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AG-221-CP-002
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetic; Healthy; Male; AG-221; [14C]; Single dose; Oral; Intravenous
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100-mg AG-221 oral solution + a microtracer of [14C]-AG- 221 (Experimental): Subjects will receive a 100 mg AG-221 to be swallowed with 240 mL of room-temperature, non-carbonated water.
  Interventions: Drug: AG-221
- 100-mg AG-221 tablet + 100 micrograms [14C] AG-221 (Experimental): Formulated tablet containing 100 mg AG-221 + IV solution containing 100 micrograms [14C] AG-221
  Interventions: Drug: AG-221; Radiation: 14C AG-221

INTERVENTIONS:
Drug: AG-221 — Part 1: oral solution containing 100 mg [14C]-AG-221
Radiation: 14C AG-221 — 5 mL of 100 micrograms [14C] AG-221 given intravenously 4 hours after swallowing the formulated tablet.
  Arms: 100-mg AG-221 tablet + 100 micrograms [14C] AG-221

SUMMARY:
This is a single-center, 2-part, open-label study to evaluate the metabolism and excretion and absolute bioavailability of [14C]-AG-221 in healthy male subjects. It is planned for 14 subjects to be enrolled; each subject will participate in a screening phase, a baseline phase, a treatment phase, and a follow up phone call. Blood, urine and fecal samples will be collected in Part 1 for analyses. Blood samples will be collected in Part 2. Subjects can only participate in either Part 1 or Part 2.

DETAILED DESCRIPTION:
This will be a single-center, open-label, 2-part study in healthy adult males (n = 14). Parts 1 and 2 may be conducted in parallel.

Each subject will participate in a screening phase, a baseline phase, a treatment phase, and a follow up phone call. Subjects who have met all inclusion criteria and none of the exclusion criteria at screening will return to the clinical site on Day 1 for baseline assessments.

Part 1: Absorption, metabolism, and excretion (AME) Approximately 8 subjects will be enrolled in Part 1. Subjects will check into the clinic on the day before dosing. Following a 10 hour overnight fast, subjects will receive a single 100-mg dose of AG-221 solution containing a microtracer of [14C] AG 221 (~ 300 nCi) under fasted conditions. The study drug will be administered as an oral solution with approximately 240 mL of room temperature, non-carbonated water.

Blood, urine, and fecal samples (and vomitus, if applicable) will be collected throughout the study for pharmacokinetic (PK), mass balance, and/or clinical laboratory assessments. Safety will be monitored throughout the study. Subjects will be discharged from the clinical site on Day 22 following completion of the required study procedures. Subjects will return to the unit on Day 29 for the last PK blood draw.

Urine and fecal samples will be collected each day until Day 22 (or the point of discharge if earlier) for measurement of total [14C] radioactivity. Blood samples for radioanalysis and PK assessment, inclusive of metabolite profiling/characterization, will be collected at pre-dose and at specified intervals through Day 29. Total [14C]-radioactivity in whole blood, plasma, urine, and feces (and vomitus, if applicable ) will be determined.

Part 2: Absolute bioavailability:

Approximately 6 subjects will be enrolled in Part 2. Qualified subjects who have met all inclusion criteria and none of the exclusion criteria at screening will return to the clinical site on Day 1, and will be housed at the clinical site from Day 1 until Day 3.

After an overnight fast of at least 10 hours, approximately 6 subjects will receive an oral dose (coated tablet) of 100 mg of AG-221 at Hour 0 on dosing day (Day 1). The study drug will be administered orally with approximately 240 mL of water. Four hours after the oral dose, the subjects will receive 100 micrograms AG-221 containing ~300 nCi of [14C]-AG-221administered as an intravenous bolus over approximately 2 minutes.

Subjects will be discharged from the unit upon completion of the 48 hour PK blood draw on Day 3. Subjects will return to the unit for additional PK blood draws on Days 5, 8, 11, 15, 18, 22, and 29.

No urine and fecal samples will be collected in Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy adult male of any race and between 18 to 55 years of age, inclusive, at the time of signing the informed consent document.
2. Understands and voluntarily signs an informed consent document before any study related assessments/procedures are conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Must practice true abstinence1 or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a female of childbearing potential (FCBP)2 while participating in the study and for at least 28 days following the last dose of Investigational Product (IP), even if he has undergone a successful vasectomy.
5. Must have a Body Mass Index (BMI) between 18 and 33 kg/m2, inclusive, at screening.
6. Must be healthy as determined by the Investigator on the basis of medical history, physical examination (PE), clinical laboratory test results, vital signs, and 12-lead Electrocardiograms (ECG) at screening:

   * Must be afebrile (febrile is defined as ≥ 38.5°C or 101.3°F)
   * Supine systolic blood pressure (BP) must be in the range of 90 to 140 mmHg, supine diastolic BP must be in the range of 50 to 90 mmHg, and pulse rate must be in the range of 40 to 110 bpm
   * Normal or clinically acceptable 12-lead ECG, with a QT interval, corrected for heart rate using the Fridericia formula (QTcF) value ≤ 430 msec

Exclusion Criteria:

1. History of any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition, including the presence of clinically significant (CS) laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study.
3. Any condition that confounds the ability to interpret data.
4. Exposed to an investigational drug (new chemical entity) within 30 days preceding dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
5. Participation in more than one other radiolabeled investigational drug study within 12 months prior to check-in (Day -1).

   Note: The previous radiolabeled investigational drug must have been received more than 6 months prior to check-in (Day -1) and the total planned exposure from this current study and the previous study must be within the recommended levels considered safe, per US CFR governing Protection of Human Subjects; radioactive drugs for certain research uses.
6. Exposure to significant radiation (eg, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check-in (Day -1).
7. Used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days of dose administration.
8. Used any nonprescription systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days of dose administration.
9. Used cytochrome P450 (CYP)3A inducers and/or inhibitors (including St. John's wort) within 30 days of dose administration. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inhibitors and/or inducers of CYP3A.
10. Received a live vaccination within 90 days of dose administration.
11. Has any surgical or medical conditions possibly affecting ADME (Absorption, distribution, metabolism, and excretion), eg, bariatric procedure, or plans to have elective or medical procedures performed during the conduct of the trial.

    Prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study.
12. Donated blood or plasma within 8 weeks before dose administration to a blood bank or blood donation center.
13. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dose administration, or positive drug screening test reflecting consumption of illicit drugs.
14. History of alcohol abuse within 2 years before dose administration, or positive alcohol screen.
15. Known to have serum hepatitis or known to be a carrier of HBsAg (Hepatitis B surface antigen) or HCV Ab (Hepatitis C viral antibody), or have a positive result to the test for HIV (Human immunodeficiency virus ) antibodies at screening.
16. Smokes more than 10 cigarettes per day, or the equivalent in other tobacco products.
17. Employed by the clinical site, or is related to an employee of the clinical site.
18. History of less than one bowel movements per day.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-05-14 (Actual); Primary Completion 2015-07-21 (Actual); Study Completion 2015-07-21 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Total [14C] Whole blood and plasma | Approximately 3 weeks
  Total [14C]-radioactivity in whole blood and plasma
Pharmacokinetics - Total [14C] urine and feces | approximately 3 weeks
  Total [14C]-radioactivity in urine, and feces (and vomitus, if applicable).
Pharmacokinetics - Total [14C] Cumulative excretion | approximately 3 weeks
  Cumulative excretion of total [14C]-radioactivity (as a fraction of the radioactive dose) in urine and feces (and vomitus, if applicable)
Pharmacokinetics - Total [14C] radioactivity | approximately 4 weeks
  Total [14C]-radioactivity whole blood-to-plasma ratios
Pharmacokinetics - Total [14C] metabolites | approximately 3 weeks
  Metabolite profiling / characterization in select plasma, urine, and fecal samples
Pharmacokinetics: Metabolite profiling and characterization in select biological matrices (Part 1) | approximately 4 weeks
  The analysis for metabolite profiles and characterization are qualitative and there are no units for the analysis.
Pharmacokinetics - Cmax | approximately 4 weeks
  Maximum observed plasma concentration
Pharmacokinetics - AUC | approximately 4 weeks
  Area under the plasma concentration-time curve
Pharmacokinetics - Tmax | approximately 4 weeks
  Time to maximum observed plasma concentration
Pharmacokinetics -T1/2 | approximately 4 weeks
  Estimate of the terminal elimination half-life

SECONDARY OUTCOMES:
Adverse Events (AEs) | approximately 8 weeks
  An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study.

CONTACTS AND LOCATIONS:
Overall Officials: Edward O'Mara, MD, Study Director — Celgene Corporation

REFERENCES:
- [Derived] Wang X, Chen J, Reyes J, Zhou S, Palmisano M, Li Y. A Phase 1, Open-Label Study in Healthy Subjects to Evaluate the Absolute Bioavailability of AG-221 by a Microtracer Approach. Oncol Ther. 2020 Jun;8(1):91-102. doi: 10.1007/s40487-019-0097-7. Epub 2019 Jul 19. PMID 32700065